CLINICAL TRIAL: NCT02582866
Title: A Multicenter, Open-label, Follow-up Study to Assess the Long-term Use of Lacosamide (Flexible Dose From 200 to 600 mg/Day) Used as Monotherapy in Subjects Who Completed SP0994 and Received Lacosamide Monotherapy Treatment
Brief Title: A Clinical Study to Investigate the Long-term Use of Lacosamide as Monotherapy in Subjects Who Completed Study SP0994
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP1042; 2015-001549-96 (EudraCT Number)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Epilepsy; Partial onset seizures; Tonic-clonic seizures; Monotherapy; AED
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Lacosamide (LCM) will be administered orally twice daily from 200 mg/day to 600 mg/day (at approximately 12 hour intervals in the morning and in the evening) in 2 divided doses. Medication must not be chewed and must be swallowed with a sufficient amount of fluid. The investigator may maintain the subject's LCM dose, decrease the dose in decrements of 100 mg/day per week to a minimum dose of LCM 200 mg/day, or increase the dose in increments of 100 mg/day per week up to a maximum dose of LCM 600 mg/day.
  Subjects stopping LCM should be tapered off LCM at recommended decreasing steps of 200 mg/day/week. A slower taper (eg, 100 mg/day/week) or faster taper is permitted, if medically necessary; however, the maximum duration of tapering should not exceed 6 weeks.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — * Pharmaceutical Form: Oral tablets
  * Concentration: 50 mg
  * Route of Administration: Oral administration
  Other Names: Vimpat; SPM927; LCM

SUMMARY:
Study is conducted to evaluate the long-term safety and tolerability of lacosamide (LCM) in patients receiving LCM in SP0994 [NCT01465997]. The study will enable collection of additional monotherapy safety data, and will facilitate access to treatment until commercial availability for monotherapy use.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board /Institutional Ethics Committee approved written Informed Consent Form (ICF) is signed and dated by the subject or by the parent(s) or legal representative. The ICF or a specific Assent form, where required, will be signed and dated by minors
* Subject/legal representative is considered reliable and capable of adhering to the protocol, visit schedule, and medication intake according to the judgment of the investigator
* Subject has completed the Termination Visit of SP0994 [NCT01465997] and has been treated with lacosamide monotherapy

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to lacosamide (LCM)
* Subject experienced a seizure at the 3rd target dose (i.e. LCM 600 mg/day) during SP0994
* Subject required another Anti Epileptic Drug (AED) for the treatment of seizures
* Subject meets a "must" withdrawal criteria for SP0994
* Subject is experiencing an ongoing Serious Adverse Event from SP0994
* Female subject who is pregnant or nursing, and/or a woman of childbearing potential who is not surgically sterile, 2 year postmenopausal or does not practice one highly effective method of contraception, unless sexually abstinent, for the duration of the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (46):
- Bulgaria (3):
  - Sp1042 805, Blagoevgrad
  - Sp1042 807, Pazardzhik
  - Sp1042 811, Sofia
- Finland (2):
  - Sp1042 205, Helsinki
  - Sp1042 207, Kuopio
- Sp1042 236, Nancy, France
- Germany (5):
  - Sp1042 263, Altenburg
  - Sp1042 265, Bad Neustadt an der Saale
  - Sp1042 269, Leipzig
  - Sp1042 256, Marburg
  - Sp1042 259, Osnabrück
- Japan (6):
  - Sp1042 831, Asaka
  - Sp1042 834, Kagoshima
  - Sp1042 844, Kamakura
  - Sp1042 835, Nagoya
  - Sp1042 837, Okayama
  - Sp1042 847, Sapporo
- Sp1042 751, Riga, Latvia
- Sp1042 547, San Luis Potosí City, Mexico
- Philippines (2):
  - Sp1042 672, Pasig
  - Sp1042 676, Quezon
- Poland (3):
  - Sp1042 340, Katowice
  - Sp1042 342, Lublin
  - Sp1042 343, Warsaw
- Romania (3):
  - Sp1042 576, Bucharest
  - Sp1042 570, Iași
  - Sp1042 572, Târgu Mureş
- Russia (6):
  - Sp1042 387, Kazan'
  - Sp1042 389, Kazan'
  - Sp1042 401, Moscow
  - Sp1042 392, Novosibirsk
  - Sp1042 397, Saint Petersburg
  - Sp1042 400, Saint Petersburg
- South Korea (4):
  - Sp1042 521, Daegu
  - Sp1042 518, Daejeon
  - Sp1042 517, Seoul
  - Sp1042 519, Seoul
- Sweden (3):
  - Sp1042 440, Gothenburg
  - Sp1042 442, Linköping
  - Sp1042 438, Stockholm
- Switzerland (3):
  - Sp1042 651, Aarau
  - Sp1042 654, Biel
  - Sp1042 653, Lugano
- Ukraine (3):
  - Sp1042 622, Chernihiv
  - Sp1042 626, Kharkiv
  - Sp1042 625, Odesa

REFERENCES:
- [Result] Ben-Menachem E, Dominguez J, Szasz J, Beller C, Howerton C, Jensen L, McClung C, Roebling R, Steiniger-Brach B. Long-term safety and tolerability of lacosamide monotherapy in patients with epilepsy: Results from a multicenter, open-label trial. Epilepsia Open. 2021 Sep;6(3):618-623. doi: 10.1002/epi4.12522. Epub 2021 Aug 2. PMID 34265173
- [Result] Inoue Y, Liao W, Wang X, Du X, Tennigkeit F, Sasamoto H, Osakabe T, Hoshii N, Yuen N, Hong Z. Safety and efficacy of adjunctive lacosamide in Chinese and Japanese adults with epilepsy and focal seizures: A long-term, open-label extension of a randomized, controlled trial. Epilepsy Res. 2021 Oct;176:106705. doi: 10.1016/j.eplepsyres.2021.106705. Epub 2021 Jun 29. PMID 34246118
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in January 2016 and concluded in January 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Lacosamide: Lacosamide (LCM) was administered orally, twice daily from 200 mg/day to 600 mg/day, in 2 divided doses at approximately 12 hour intervals in the morning and in the evening. The investigator may have maintained the subject's LCM dose, decreased the dose in decrements of 100 mg/day per week to a minimum dose of LCM 200 mg/day, or increased the dose in increments of 100 mg/day per week up to a maximum dose of LCM 600 mg/day.
  Participants stopping LCM should have been tapered off LCM at recommended decreasing steps of 200 mg/day/week. A slower taper (eg, 100 mg/day/week) or faster taper was permitted but the duration of tapering should not have exceeded 6 weeks.
Period: Overall Study
Arm/Group | Lacosamide
Started | 106
Completed | 84
Not Completed | 22
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 7
Not completed — Investigator decision | 5
Not completed — Participant wants to get pregnant | 1
Not completed — Pregnancy | 2
Not completed — Sponsor decision | 1
Not completed — Withdrawal due to personal reasons | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all study participants in the Enrolled Set (ES) who received at least 1 dose of study medication in SP1042.
Arm/Group | Lacosamide
Number analyzed (Participants) | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 90
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 19
  White | 86
  Other/Mixed | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Adverse Events (AEs) Reported Spontaneously by the Subject and/or Caregiver or Observed by Investigator
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE could, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study medication.
Time Frame: From Visit 1 (Week 0) to Final Visit (up to Week 158)
Population: The SS consisted of all study participants in the ES who received at least 1 dose of study medication in SP1042.
Measure: Number; unit: percentage of participants
Groups:
- Lacosamide (SS): Lacosamide (LCM) was administered orally, twice daily from 200 mg/day to 600 mg/day, in 2 divided doses at approximately 12 hour intervals in the morning and in the evening. The investigator may have maintained the subject's LCM dose, decreased the dose in decrements of 100 mg/day per week to a minimum dose of LCM 200 mg/day, or increased the dose in increments of 100 mg/day per week up to a maximum dose of LCM 600 mg/day.
  Participants stopping LCM should have been tapered off LCM at recommended decreasing steps of 200 mg/day/week. A slower taper (eg, 100 mg/day/week) or faster taper was permitted but the duration of tapering should not have exceeded 6 weeks.
  Participants formed the Safety Set (SS).
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 106
percentage of participants | 59.4

2. Primary Outcome: Percentage of Participants That Withdrew Due to Adverse Events (AEs)
Description: as for outcome 1
Time Frame: From Visit 1 (Week 0) to Final Visit (up to Week 158)
Population: The SS consisted of all study participants in the ES who received at least 1 dose of study medication in SP1042.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 106
percentage of participants | 0.9

3. Primary Outcome: Percentage of Participants Experiencing Any Serious Adverse Events (SAEs) Reported Spontaneously by the Subject and/or Caregiver or Observed by Investigator
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the study participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Visit 1 (Week 0) to Final Visit (up to Week 158)
Population: The SS consisted of all study participants in the ES who received at least 1 dose of study medication in SP1042.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 106
percentage of participants | 14.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 (Week 0) to Final Visit (up to Week 158)
Arm/Group | Lacosamide (SS)
All-Cause Mortality (participants affected / at risk) | 1/106
Serious Adverse Events (participants affected / at risk) | 15/106
Other Adverse Events (participants affected / at risk) | 19/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=106)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1)
Device Dislocation (General disorders) | 1 (1)
Sudden Unexplained Death In Epilepsy (General disorders) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1)
Post Gastric Surgery Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arteriogram Coronary (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2)
Ischaemic Stroke (Nervous system disorders) | 1 (1)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=106)
Nasopharyngitis (Infections and infestations) | 8 (17)
Headache (Nervous system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02582866/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT02582866/SAP_001.pdf